CLINICAL TRIAL: NCT05779800
Title: Clinical Comparison of the Use of Flowable Resin Composite Stent Versus Periodontal Pack to Reduce Donor Site Morbidity After Free Gingival Graft Harvesting: A Randomized Clinical Trial
Brief Title: The Use of Flowable Resin Composite Stent in Reduction of Donor Site Morbidity After Free Gingival Graft Harvesting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Elsayed Ahmed Hassan Temraz, demonstrator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9322
Record Dates: First submitted 2023-02-25; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Free Gingival Graft
Keywords: palatal donor site; Gingival Recession; Periodontal Diseases; Protective Agents; flowable composite
MeSH Terms: conditions — Gingival Recession; Periodontal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flowable resin composite stent group (Experimental): Flowable resin composite is a bio compatible material used in dental field many years ago.
  Interventions: Device: Flowble resin composite stent
- Periodontal pack group (Active Comparator): Non eugenol containing periodontal pack used in periodontal surgeries to protect the wound.
  Other name :COE_PAK
  Interventions: Device: periodontal pack

INTERVENTIONS:
Device: Flowble resin composite stent — Flowble resin composite is a filling material used in operative dentistry and characterized by being flow and easily adapting the surfaces.
  Other Names: NEXOCOMP FLOW
  Arms: Flowable resin composite stent group
Device: periodontal pack — Non eugenol containing dressing supplied in two tubes
  Other Names: COE-PAK
  Arms: Periodontal pack group

SUMMARY:
After harvesting free gingival graft from the hard palate, Postoperative pain as well as bleeding are the most common complications.Different agents were used to protect the denuded areas on the palate as gelatin sponge, Hyaluronic acid gel and platelet rich fibrin (PRF) but still no gold standard material is present.

PICO format:

P: patients with mucogingival problems in need for free gingival graft or de-epithelialized connective tissue graft.I: Flowable resin composite stent. C: Periodontal pack. O: Post-operative pain T: day 3, 7, 14, 21 and 42 postoperative.

Aim of the study:

To compare the effect of flowable composite stent versus periodontal pack applied to palatal donor site after free gingival graft harvesting in terms of post-operative pain reduction.

DETAILED DESCRIPTION:
Intervention:

Flowable resin composite stent.

Procedure:

After the palatal sites be anaesthetized with 0.3 ml of a solution of 4% Articaine and 0.001% Adrenalin. Graft harvesting will be performed by basic surgical techniques described by Miller (1982). A rectangular shaped piece of mucosa will be harvested from the area of the hard palate by a split-thickness dissection.

The graft will then be used as it on the recipient bed. The graft dimensions will be recorded (width and length).

Denuded palatal area will then be protected using one of the following options:

1. Periodontal pack (control group)
2. flowble resin composite NEXOCOMP FLOW (intervention group)

Postoperative instructions:

Postoperative instructions will include discontinuing tooth brushing and flossing around the surgical sites until the day of periodontal dressing removal (day 7).

Patients will be directed to consume only soft foods during the first week and to avoid any mechanical trauma.

Patients will be scheduled to be seen on days 7, 14, 21 and 42 Periodontal pack and flowble resin composite stent will be first removed on day 7, and donor sites will be evaluated using selected parameters in both groups.

Thereafter, all patients will be followed up on days 14, 21 and 42 for further evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mucogingival defects scheduled for free gingival graft or de-epithelialized connective tissue graft.
* Systemically healthy

Exclusion Criteria:

* Smokers
* Occlusal trauma at site of graft
* Pregnancy and lactation
* Patients allergic to the used agents
* Severe gagging reflex

Ages: 21 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2023-11-08 (Estimated); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | on day 7
  Pain score reported by the patient directly through Visual Analogue Scale score (between 0 and 100. 0: no pain, 10: minimal pain, 50:moderate pain, 100: severe pain)

SECONDARY OUTCOMES:
Color match | On day 42
  The color of the palatal mucosa will be assessed by comparing it with that of the adjacent and opposite side by using the objective VAS (VAS score 0-10) represented by a continuous line, by a clinician blinded to the treatment group assignment.
wound size | at day 21
  To be recorded using (UNC 15) periodontal probe to the nearest measurement of 0.5 mm , length and width only

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Cairo univesity, Cairo, Manial, Egypt